CLINICAL TRIAL: NCT06280014
Title: Evaluation of the Effects of Mefenamic Acid and Dexketoprofen on Postoperative Pain, Edema and Trismus in Impacted Wisdom Dental Surgery
Brief Title: Evaluation of the Effects of Mefenamic Acid and Dexketoprofen on Postoperative Wisdom Dental Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor Serap Keskin Tunc, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: YYU-09/15.12.2021
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Tooth, Impacted; Tooth Diseases
Keywords: impacted wisdom teeth; dexketoprofen; mefenamic acid
MeSH Terms: conditions — Tooth, Impacted; Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mefenamic acid was used to see post operative effects after extraction of 3rd molar in study group (Experimental): In this study of 30 patients, 22 females and 8 males, 60 fully impacted lower wisdom teeth were extracted bilaterally and in the same position. One of the bilaretal teeth of the patients was randomly selected and mefenamic acid was used as a drug to see post operative effects after extraction of impacted 3rd molars in the study group.
  Interventions: Procedure: Surgery of impacted mandibular wisdom teeth
- Dexketoprofen was used to see post operative effects after extraction of 3rd molar in control group (Placebo Comparator): Bilateral impacted wisdom teeth of the patients were randomly selected. After the tooth in the experimental group was extracted, the other impacted wisdom tooth was selected as the control group and dexketoprofen was used as a drug to see post operative effects.
  Interventions: Procedure: Surgery of impacted mandibular wisdom teeth

INTERVENTIONS:
Procedure: Surgery of impacted mandibular wisdom teeth — All surgical procedures were performed by the same surgeon using the standard surgical technique described below. The anesthetic used was 4% articaine with 1:100,000 adrenaline. In all patients, a sulcus incision was made in the lower second molar and an envelope incision in the third molar region, the mucoperiosteal flap was removed, and extraction was performed with a bone elevator and a third molar elevator. If necessary, the impacted molar was incised with a high-speed dental handpiece and a fissure bur. The wound was irrigated with copious amounts of saline, and the wound edges were carefully sutured with simple 4.0 silk braided non-absorbable sutures. After extraction of impacted wisdom tooth, the patient was given mefenamic acid as a medication.
  Other Names: Surgery of impacted molar teeth
  Arms: Mefenamic acid was used to see post operative effects after extraction of 3rd molar in study group
Procedure: Surgery of impacted mandibular wisdom teeth — All surgical procedures were performed by the same surgeon using the standard surgical technique described below. The anesthetic used was 4% articaine with 1:100,000 adrenaline. In all patients, a sulcus incision was made in the lower second molar and an envelope incision in the third molar region, the mucoperiosteal flap was removed, and extraction was performed with a bone elevator and a third molar elevator. If necessary, the impacted molar was incised with a high-speed dental handpiece and a fissure bur. The wound was irrigated with copious amounts of saline, and the wound edges were carefully sutured with simple 4.0 silk braided non-absorbable sutures. After extraction of impacted wisdom tooth, the patient was dexketoprofen as a medication.
  Other Names: Surgery of impacted molar teeth
  Arms: Dexketoprofen was used to see post operative effects after extraction of 3rd molar in control group

SUMMARY:
This study was administered to 22 female and 8 male patients. Patients with impacted wisdom teeth on both sides of the mandible were selected. After impacted tooth extraction, the patient used mefenamic acid on one side and dexketoprofen on the other side for postoperative pain relief. The effects of these two materials on patient comfort were investigated.

DETAILED DESCRIPTION:
The aim of this study; to compare the effects of dexketoprofen and mefanamic acid on pain, edema and trismus after lower impacted wisdom teeth surgery. 60 impacted wisdom teeth in 30 healthy individuals who applied to Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery with an indication for extraction of impacted lower wisdom teeth were included in the study. 60 impacted wisdom teeth belonging to individuals were randomly divided into two groups (A and B). In a randomized, controlled, double-blind study, dexketoprofen (A) and mefanamic acid (B) were given to patients immediately after surgery. VAS (Visual Analog Scale) was used for pain assessment and assessment was made at 3, 6, 12 and 24 hours and 2, 3, 4, 5, 6 and 7 days. For the evaluation of edema, the facial measurements of the patients before the operation were recorded and repeated on the 2nd and 7th postoperative days. Preoperative maximum mouth opening measurement for trismus assessment was repeated on the 2nd and 7th postoperative days and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with bilateral fully impacted mandibular wisdom teeth

Exclusion Criteria:

* Patients were excluded from the study if they did not understand the clinical procedures of the study,
* Had allergies or intolerance to any of the substances used in the study,
* Patients on anticoagulant or psychiatric treatment,
* Pregnant or breastfeeding,
* Patients using oral contraceptiveswere,
* Diabetic,
* Patients with periodontal disease or active infection,
* Poor oral hygiene

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Mouth opening measurements | 0-28 days
  The distance between the incisals of the patient's central teeth at maximal mouth opening.
Facial edema | 0-28 days
  Measurement between facial craniometric points (angulus-tragus, angulus-lateral canthus, angulus-nasal base, angulus-lateral canthus, and angulus-pogonion). The number of participants in the split mouth model was 22. A total of 44 impacted teeth were extracted and edema was measured before and 1 week after each extraction.
Visual Analog Scale | 0-28 days
  A numerical rating scale VAS was used for pain analysis (0=no pain, 10=most severe pain). The pain levels at 24 hours, 48 hours and 1 week after the surgical procedure were recorded on the patient follow-up form by all patients who participated in the study by explaining that there was no pain at the "zero" level and the most severe pain known at the "10" level on the pain scale, which was organized as a 10 cm horizontal line on the prepared forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Serap Keskin Tunc, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided